CLINICAL TRIAL: NCT03795337
Title: Hypofractionated Radiosurgery for Localised Prostate Cancer
Brief Title: Hypofractionated Radiosurgery for Localised Prostate Cancer (HYPOSTAT-II)
Acronym: HYPOSTAT-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Luebeck (Other); Saphir Radiosurgery Center Northern Germany (Unknown)
Responsible Party: Principal Investigator, Juergen Dunst, Prof., Clinical Professor, Director, Head of Department, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZKS-121-08; ARO-2018-4 (Other: German Cancer Society)
Record Dates: First submitted 2018-12-19; First posted 2019-01-07 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: Hypofractionation; Prostate Cancer; Radiotherapy; long-term toxicity
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated Radiosurgery (Experimental): 5 fractions with 7 Gy, total dose 35 Gy
  Interventions: Radiation: Hypofractionated Radiosurgery

INTERVENTIONS:
Radiation: Hypofractionated Radiosurgery — Image-guided stereotactic Linac based RT preferable with "dedicated radiosurgery system" such as CyberKnife

SUMMARY:
Hypofractionated radiosurgery has been investigated in a few trials and appears to be safe and feasible.

Investigators initiated this multicenter phase II prospective trial to analyse feasibility (toxicity) of hypofractionated radiosurgery with 5 fractions in patients with localised prostate cancer under the hypothesis that the ratio of patients with late toxicity ≥ grade 2 after 3 years amounts 4.1% and is significant lower than 12.3% and 8.7% currently.

DETAILED DESCRIPTION:
Experimental radiosurgery of prostate with 5 fractions each with 7,00 Gy (total application rate of 35,00 Gy).

Planned visits are: Baseline, visits at every radiation day and eight follow ups (4-6 weeks, 3 months, 6 months, 1 year and every year thereafter after last day of radiation).

ELIGIBILITY:
Inclusion Criteria:

* non-metastatic, histopathologically confirmed prostate carcinoma cT 1-3 N0 M0
* Gleason-grade ≤7
* Guideline-based staging
* Age ≥ 60 years
* PSA < 15 ng / ml
* Volume of the prostate < 80 cm³
* IPSS-Score ≤ 12
* Written informed consent

Exclusion Criteria:

* Age ≤ 60 years
* History of prior pelvic radiotherapy
* Contraindication to MRI or Fiducial marker implantation (e.g. allergy to gold),
* Immunosuppressive therapy
* Relevant comorbidity thought to adversely affect treatment compliance,
* Legal incapacity or lack of informed consent

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 475 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Late toxicity measured with Radiation Therapy Oncology Group-(RTOG)-Score | 3, 6-9, 12-15 months and thereafter annually for 4 years after radiotherapy

SECONDARY OUTCOMES:
Acute toxicity analysed by Adverse Event (AE)- and Serious Adverse Event (SAE)-reports. | 4-6 weeks after radiotherapy; 3, 6-9, 12-15 months after radiotherapy thereafter annually for 4 years after radiotherapy
Prostate Specific Antigen (PSA) | At the time of inclusion; 4-6 weeks after radiotherapy; 3, 6-9, 12-15 months after radiotherapy thereafter annually for 4 years after radiotherapy
International Prostate Symptom Score (IPSS) | At the time of inclusion; 4-6 weeks after radiotherapy; 3, 6-9, 12-15 months after radiotherapy thereafter annually for 4 years after radiotherapy
EORTC Quality of Life Questionnaire (QLQ) C30 | At the time of inclusion; 12-15 months after radiotherapy thereafter annually for 4 years after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Dunst, Prof., Principal Investigator — University Hospital Schleswig-Holstein; Alexander Muacevic, Prof., Principal Investigator — European CyberKnife Center Munich
Locations (8):
- Germany (8):
  - Charité Berlin, Department of Radiation Oncology and Radiotherapy (CVK), Berlin
  - University Medical Center Cologne, Department of Radiation Oncology, Cyberknife- and Radiotherapy, Cologne
  - CyberKnife Centrum Mitteldeutschland, Erfurt
  - Saphir Radiosurgery Center Frankfurt am Main, Frankfurt am Main
  - University Hospital Frankfurt, Department of Radiation Therapy and Oncology, Frankfurt am Main
  - Saphir Radiosurgery Center Northern Germany, Kiel
  - University Medical Center Schleswig-Holstein, Kiel
  - European Cyberknife Center Munich, Munich